CLINICAL TRIAL: NCT05367011
Title: Etude de Cohorte de Suivi thérapeutique de l'antibiothérapie Chez Les Patients de réanimation
Brief Title: Therapeutic Monitoring of Antibiotics in Intensive Care Patients: a Cohort Study PopTDM-ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PopTDM-ICU
Record Dates: First submitted 2022-03-18; First posted 2022-05-10 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-05

CONDITIONS: Intensive Care Unit; Antibiotic Therapy; Pharmacokinetic
Keywords: Antibiotic; Intensive care; Therapeutic drug monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intensive care patients are exposed to serious infections. Mortality linked to these infections remains high and antibiotic therapy treatment optimization is one of the key points of therapeutic success . Pharmacokinetic therapeutic monitoring and dosage adjustments are recommended for large families of antibiotics such as glycopeptides and aminoglycosides for a long time, but to this day still insufficiently practiced. Concerning Beta-Lactamines this practice is recommended by french society of pharmacology and therapeutic (SFPT) and french society of anesthesiology and intensive care (SFAR) since 2018.

The main goal of the POP-TDM-ICU study is to find the predictive factors of clinical therapeutic efficacy of antibiotic therapy in sepsis or septic shock in intensive care, among which the use of the dosage pharmacokinetics of antibiotic therapy (TDM = Therapeutic Drug Monitoring).

This study is a non-interventional study. Patients bacterial samples already collected in standard care and additional plasma samples will be collected as part of a biological collection with the consent of the patient or family member.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 year-old.
* Patient hospitalized in intensive care,
* Patient receiving an antibiotic for sepsis or septic shock
* Patient or family member who does not object to participating in the study

Exclusion Criteria:

Patient at risk of death, for a cause other than infectious, within 48 hours following the introduction of antibiotic therapy.

* Patient receiving antibiotic treatment for antibiotic prophylaxis.
* Patients benefiting from enhanced protection, namely: minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social establishment, adults under legal protection.
* Pregnant and / or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients with to serious infections
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical therapeutic efficacy at the end treatment or at day 14 in the event of prolonged treatment, defined by the combination of the following 3 points. | up to 14 days
  * A disappearance of all signs and symptoms of infection, or a marked decrease in the severity of infection defined by evolution of Sequential Organ Failure Assessment (SOFA) Score. SOFA score describes the time course of multiple organ dysfunction using a limited number of routinely measured variables. The function of six organ systems is scored from 0 (no organ dysfunction) to 4 (severe organ dysfunction), and the individual organ scores are then summed to a total score between 0 and 24.
  * Absence of necessary therapeutic escalation during the duration of treatment
  * No antibiotic treatment for the same pathology within 48 hours of stopping treatment.